CLINICAL TRIAL: NCT05645367
Title: Associations of Lipid Measures With Premature Myocardial Infarction: a Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Yue LI (Other)
Responsible Party: Sponsor-Investigator, Yue LI, Professor, First Affiliated Hospital of Harbin Medical University
Organization: First Affiliated Hospital of Harbin Medical University (Other)
Other Study IDs: lipid and PMI
Record Dates: First submitted 2022-12-02; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Lipid Disorder; Premature Myocardial Infarction
MeSH Terms: conditions — Lipid Metabolism Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- premature myocardial infarction: AMI with onset age less than 55 years for men and 65 years for women.
  Interventions: Other: No intervention
- control: AMI with onset age not less than 55 years for men and 65 years for women.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a post-hoc analysis of a cross-sectional study.

SUMMARY:
Acute myocardial infarction (AMI) is the first cardiovascular cause of death that seriously threatens human health worldwide. Its incidence rate and mortality are increasing year by year and becoming younger. According to statistics, the average age of men and women with AMI for the first time is 65.6 years old and 72 years old respectively, of which 4%~10% AMI occurred before 45 years old. At present, there is no uniform age threshold for young AMI. Generally speaking, AMI with onset age less than 55 years for men and 65 years for women is called early-onset AMI, accounting for 5%~13% of AMI. Compared with elderly patients with AMI, patients with early onset AMI have different risk factors, clinical characteristics and prognosis, such as lower proportion of patients with diabetes and hypertension, more single vessel lesions and rare left main artery involvement, and higher long-term recurrence rate and mortality. Although the progress of preventive measures and treatment methods has reduced the hospitalization rate of elderly AMI patients, the number of young AMI patients in hospital is still rising. Therefore, in-depth analysis of the characteristics of risk factors of early onset AMI and early intervention are of great significance to reduce the risk of onset and improve long-term prognosis.

Hyperlipidemia is an independent risk factor for coronary heart disease at all ages, and is more closely related to early onset AMI. It is reported that more than 50% of early onset AMI patients are accompanied by hyperlipidemia. However, at present, the research on the relationship between blood lipids and early onset AMI is limited to the comparison of the level of single lipid component between early onset AMI and different control groups, or the comparative analysis of the relationship between a specific lipid component and the risk of early onset AMI with young healthy people. There is no research to compare the correlation between various lipid components and the risk of early onset AMI. Therefore, this study plans to deeply analyze the correlation between different blood lipid components and their ratios and early onset AMI, and further analyze which blood lipid indicators are most closely related to early onset AMI through large sample clinical research data, taking late onset AMI patients as the control, which should be paid early attention to and strictly managed.

ELIGIBILITY:
Inclusion Criteria:

* According to the fourth Universal Definition of Myocardial Infarction (2018), the clinical diagnosis was acute myocardial infarction (AMI), including type 1, 2, 3, 4b and 4c.
* Complete coronary angiography
* Complete biochemical and blood lipid tests

Exclusion Criteria:

* Recurrent AMI
* The onset of AMI exceeds 7 days
* Continuous taking of lipid-lowering drugs ≥ 5 days
* Patients with missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AMI patients who completed coronary angiography in the First Affiliated Hospital of Harbin Medical University from September 1, 2021 to September 31, 2022 were included consecutively to establish an AMI research queue. Baseline information such as demographic information, medical history information and laboratory examination results were collected through the electronic medical record system.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The correlation between different blood lipid components and early onset AMI. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China